CLINICAL TRIAL: NCT04982679
Title: Relationship Between The Quadriceps Muscle Stiffness And Patellar Alignment For Healthy People
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: 20038261r
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-07

CONDITIONS: Patellofemoral Maltracking
Keywords: muscle stiffness; patellofemoral alignment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patellofemoral pain is a common disease, and it often couples with patellar malalignment. Previously, imbalance of the different quadriceps muscle heads was believed to be a causative factor of patellar malignment. However, findings from electromyography studies on quadriceps activities and patellar alignment in the last two decades were inconsistent. In order to better understand the relationship between quadriceps muscle imbalance and patellar malalignment, shear wave elastography (SWE), which can measure the passive and active muscle stiffness, may shed some new lights to this area. This study aims to examine whether the quadriceps muscle stiffness can predict the patellar position. The healthy young adult will be recruited in this study. Active and passive quadriceps muscle stiffness will be measured with the SWE in different conditions and the result will be correlated with the patellar position measured with magnetic resonance imaging (MRI). Also, electromyography (EMG) activity will be measured during the active stiffness measurement so as to establish the level of agreement between the EMG and SWE data. Linear regression will be used to calculate the relationship between different factors. The total number of subjects needed will be 55 by setting an effect size of 0.15 with two predictors, 80% power, and α at 0.05 in the linear regression.

This project will be conducted at PolyU campus and an MRI clinic in Hong Kong. Hopefully, it could be started in July 2021 and will last for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and in the range between 18 and 45 years.

Exclusion Criteria:

* Knee pain in the last 3 months;
* Previous history of knee surgery;
* People with contraindications to having MRI scanning.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subject without patellofemoral joint problem
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Patellofemoral Joint Alignment measured by MRI scanning | Within 1 hour
  Patellar displacement, patellar Alta/Baja and patellar tilt angle
Muscle stiffness measured by ultragraph using shear wave elastography | Within 1 hour
  Raw data of vastus lateralis, rectus femoris and vastus medialis obliquus shear modulus

SECONDARY OUTCOMES:
Muscle activity measured by electromyography | Within 1 hour
  EMG data of vastus lateralis, rectus femoris and vastus medialis obliquus
Muscle strength | Within 0.5 hour
  Maximum isometric knee extensor muscle strength at specific joint angle (30 degrees and 60 degrees knee flexion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hung Hom, Hong Kong